CLINICAL TRIAL: NCT01798797
Title: Integrated Diagnostic for Heart Failure
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: TRIAGE-HF
Record Dates: First submitted 2013-02-14; First posted 2013-02-26 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; HFRS; OptiVol; ICD; CRT-D
MeSH Terms: conditions — Heart Failure; Hemorrhagic Fever with Renal Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: non-randomized, all subjects who have been implanted with an ICD or CRT-D for at least 3 months

SUMMARY:
A prospective post-market study to evaluate the performance and clinic usability of heart failure risk status (HFRS) feature on CareLink.

DETAILED DESCRIPTION:
Patients with systolic heart failure (HF) implanted with Medtronic wireless implantable cardiac defibrillator (ICD) or cardiac resynchronization therapy device with defibrillation capabilities (CRT-D) devices will be enrolled in the study. The purpose of the study is to evaluate the usability of CareLink HFRS to manage a patient's heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient ( or patient's legally authorized representative) is willing and able to provide written informed consent
* Patient is willing and able to comply with the required study follow up visits
* Patient is implanted with a Medtronic wireless ICD or CRT-D device capable of OptiVol fluid monitoring feature
* Patient is on Medtronic CareLink network or is willing to be enrolled on the CareLink network
* Patient is being managed, or has been managed, by a HF clinician
* Patient has signed an informed consent for CareLink Network Services
* Patient is implanted with device for at least three months
* Patient is willing and able to transmit data using the CareLink home monitor (2490C).

Exclusion Criteria:

* Patient is participating in another study that may interfere with TRIAGE-HF protocol required procedures
* Patient with an implantable cardiac device that is indicated to reach ERI in less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with heart failure who have been implanted with an ICD or a CRT-D wirless device for at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Heart Failure Risk Status Performance Characterization | from baseline until a subject completes 8 months of follow up
  The clinical signs and symptoms of worsening HF that are associated with an Heart Failure Risk Status triggered by an OptiVol alert

SECONDARY OUTCOMES:
Heart Failure Risk Status and medical management | from baseline for each subject until they complete 8 months of follow up
  The correlation between HFRS burden and clinician's assessment of a subject risk and the subject's medical management

CONTACTS AND LOCATIONS:
Overall Officials: Sean Virani, MD, Principal Investigator — Vancouver General Hospital, Vancouver, British Columbia, Canada
Locations (3):
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Southlake Regional Health Centre, Newmarket, Ontario

IPD SHARING:
Plan to Share IPD: No